CLINICAL TRIAL: NCT01407575
Title: Buprenorphine For Treatment Resistant Depression
Acronym: BUP-TRD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Jordan F. Karp, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BUP-TRD
Record Dates: First submitted 2011-07-29; First posted 2011-08-02 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Depression; Depressive Disorder; Depressive Disorder, Major
Keywords: Buprenorphine; Receptors, opioid; Receptors, opioid, kappa
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buprenorphine (Experimental): 0.2 to 1.6mg of buprenorphine sublingual over the course of 8 weeks
  Interventions: Drug: Buprenorphine
- Placebo (Placebo Comparator): matching placebo- sublingual- over the course of 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buprenorphine — low-dose buprenorphine (range 0.2 mg/day -- 1.6 mg/day)
  Other Names: suboxone; buprenex; temgesic; subutex
  Arms: Buprenorphine
Drug: Placebo — matched placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety and efficacy of buprenorphine with placebo for adults with treatment resistant depression (TRD).

DETAILED DESCRIPTION:
Rates of treatment resistant depression (TRD) in randomized controlled trials range from 50-80% using SSRIs and SNRIs. Innovative treatments are sorely needed. Modulation of the opiate system may be a novel treatment approach for TRD. Buprenorphine (BUP) is a partial agonist at mu-receptors, and also displays affinity for kappa and delta receptors. BUP has a favorable safety profile with low risk of respiratory depression, and the pharmacokinetics are not affected by advanced age or renal dysfunction. This combination of mu-agonism and kappa-antagonism produces less dysphoria than methadone, and animal studies suggest that kappa-antagonism may exert antidepressant effects. In this small proof of concept RCT (n=20), the investigators hypothesize that there will be differences between the group receiving buprenorphine and the group receiving placebo for the following: 1) depression, anxiety, and sleep, and 2)activation of the limbic system and brain structures rich in opiate receptors and critical to reward circuits. In addition, the investigators hypothesize that there will not be differences for measures of safety (vital signs, measures of memory and reaction time, and falls) between the two groups. This pilot project will provide compelling preliminary data to support a R01 application to test the efficacy of buprenorphine for these therapeutically challenging patients.

Specific Aims:

1. Describe the relative safety of BUP in adults with TRD. The investigators hypothesize that there will be no differences in vital signs, measures of memory and reaction time, or falls between the two groups.
2. Describe the clinical effect of BUP in adults with TRD. The investigators hypothesize that depression, anxiety, sleep, and health-related quality of life, will improve to a greater extent among those receiving BUP.
3. Characterize the change in the phMRI responses to buprenorphine compared to placebo. The investigators will compare activation of the limbic system (rACC, insula, and amygdala) and brain structures rich in opiate receptors (periaqueductal grey) and critical to reward circuits (nucleus accumbens) before and immediately after administration of BUP or placebo.

The investigators are recruiting 20 community-dwelling adults, age 21 and older, who have tried at least two FDA-approved antidepressant medications at therapeutic doses each for at least 6 weeks during this episode of depression, and are still depressed.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and older
* Major depressive disorder
* Non-responder to at least 2 FDA-approved antidepressants prescribed at a therapeutic dose, each for at least 6 weeks, or is a depression non-responder from an ongoing study of late-life depression at our research clinic.
* For women of child-bearing age, must have negative pregnancy test and agree not to get pregnant while participating.

Exclusion Criteria:

* Concomitant use of strong or moderate CYP3A4 inhibitor.
* Refusal to stop all opioids.
* Refusal to discontinue all alcohol.
* Refusal to discontinue benzodiazepines other than the equivalent of lorazepam 2 mg/day prescribed at a stable dose for at least the past 2 weeks.
* Hepatic impairment (AST/ALT > 1.5 times upper normal).
* Lung disease requiring supplemental oxygen (CPAP for sleep apnea is acceptable).
* Estimated creatinine clearance <30 mL/min.
* Inability to provide informed consent.
* Depressive symptoms not severe enough (i.e., MADRS < 10) at the baseline assessment.
* Dementia, as defined by MMSE < 24 and clinical evidence of dementia
* Lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms.
* Abuse of or dependence on alcohol or other substances within the past 3 months.
* Meets criteria for history of abuse or dependence upon opioids.
* High risk for suicide.
* Contraindication to buprenorphine.
* Inability to communicate in English.
* Non-correctable clinically significant sensory impairment.
* Unstable medical illness.
* Subjects taking psychotropic medications that cannot be safely tapered and discontinued prior to study initiation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan F Karp, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buprenorphine | Placebo
Started | 7 | 6
Completed | 5 | 5
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.92 (15.88) | 64.59 (5.01) | 59.66 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale
Description: measure of depression severity Theoretical Range 0-60 lower values represent better outcome
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 33.8 (10.96) | 32.6 (2.07)

2. Primary Outcome: Blood Pressure
Description: Measure of systolic and diastolic blood pressure. 140/90 or lower is considered normal and indicates a better outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 5 | 5
mm Hg
  Systolic Blood Pressure | 138.4 (22.71) | 117.2 (28.1)
  Diastolic Blood Pressure | 91 (14.92) | 71 (15.92)

3. Primary Outcome: UKU Side Effect Rating Scale
Description: measure of side effects 46 items with scores of 0,1,2,3 possible. Theoretical range 0-138 Lower scores indicate fewer side effects
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 29.2 (13.74) | 20.2 (5.36)

4. Secondary Outcome: Brief Symptom Inventory -- Anxiety Subscale
Description: measure of anxiety Lower numbers indicate better outcome Theoretical Range 0-2.4
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 1.43 (1.1) | 0.97 (0.74)

5. Secondary Outcome: Positive and Negative Affect Scale
Description: Positive Affect Score: Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Score: Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Time Frame: 6 weeks
Population: reduced sample size verified. This was secondary to administrative error.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 4 | 4
units on a scale
  PANAS positive affect subscale | 13.75 (0.96) | 16.25 (2.99)
  PANAS negative affect subscale | 22 (11.4) | 20.5 (1.73)

6. Primary Outcome: Heart Rate
Description: Heart Rate (Beats per minute) 60-100 beats per minute is considered normal lower heart rate represent healthier outcome
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 5 | 5
Beats per minute | 87.25 (12.84) | 72.6 (19.73)

7. Primary Outcome: Weight
Description: Participant weight
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 5 | 5
lbs | 191.7 (30.02) | 203.7 (12.99)

ADVERSE EVENTS:
Arm/Group | Buprenorphine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No